CLINICAL TRIAL: NCT04726358
Title: ProCaLung - Project on Cancer of the Lung : A National Radiotherapy Quality Assurance for Stage III NSCLC
Brief Title: ProCaLung: Project on Cancer of the Lung
Acronym: ProCaLung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Collaborators: Belgian Federal Public Service, Food Chain Safety and Environment (Other Government); Belgian Cancer Registry (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-42
Record Dates: First submitted 2020-09-29; First posted 2021-01-27 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2022-09

CONDITIONS: Locally Advanced Lung Carcinoma
Keywords: NSCLC; Radiation therapy; Mediastinal adenopathy; Quality assurance; Delineation; National registry

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ProCaLung is a national registry collecting radiation treatment parameters of patients having lung cancer that extends to mediastinal lymph nodes. The project includes a peer review activity.

The purpose of this public health program is similar to an audit whose objective is to promote quality of radiation oncology in Belgium. It is run by Institut Jules Bordet on behalf of the College of Physicians for Radiotherapy Centers of the Belgian Health Federal Public Service, in close collaboration with the Belgian Cancer Registry.

All Belgian radiotherapy centers are invited to participate in ProCaLung but their participation is not mandatory. The centers who accept to participate show a commitment to quality assurance as the radiotherapy-treatment-related parameters they generate will be analyzed to establish national statistics. It includes a peer-review process based on international guidelines for mediastinal nodes delineations given for informational purposes. The public interest program also collects technical parameters as they were planned and delivered during the course of chest radiation treatment. This includes the delineations of tumors, nodes and chest organs on simulation-CT images, PET/CT images, chest-CT images and the clinical information related to the lung cancer. Results/statistics will be published at the end of the project.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC only
* Locally advanced disease (Stage III) with positive mediastinal nodes
* PET/CT staged
* Curative intent radiotherapy
* Chemotherapy (ChT): Without, Sequential ChT - Radiotherapy (RT) (max 2 cycles), Concurrent (± induction ChT)
* Prescription dose ≥ 60 Gy (EQD2)

Exclusion Criteria:

* Prior history of thoracic RT
* Malignant pleural effusion
* History of malignancy in the last 3 years, except basal-cell skin cancer and intra-epithelial neoplasia
* Progression after induction chemotherapy
* Use of concurrent targeted, immunomodulating or anti-angiogenic agents except if the patient is included in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with thoracic radiotherapy in Belgium for NSCLC with at least one positive mediastinal node.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
descriptive statistics for quality assurance (no sample size needed) | 1 year
  * Dosimetry [Non-inferiority, comparison of groups by final review group]: Mean Lung Dose, Lung V20Gy, Lung V30Gy, Mean Heart Dose, Esophagus V60Gy.
  * Waiting times, use of contrast-enhanced CT, ITV, overall treatment time, proportion of treatments with recommended organs at risk delineated, radiological treatment completion rate, chemotherapy (and immunotherapy) completion rate, use of static/rotational intensity modulation, availability of data in the electronic health record.
descriptive statistics for QA (no sample size needed) | 2 years
  * Waiting times, use of contrast-enhanced CT, ITV, overall treatment time, proportion of treatments with recommended organs at risk delineated, radiological treatment completion rate, chemotherapy (and immunotherapy) completion rate, use of static/rotational intensity modulation, availability of data in the electronic health record.

SECONDARY OUTCOMES:
Secondary endpoints related to standardization | 1 year
  * [Superiority, basis of sample size calculation] CTVn Hausdorff distance 95th percentile (HD95p) > 3mm, calculated between the initial contour of the radiotherapy (RT) center and ProCaLung's review for start and end cohorts.
  * Proportion of treatments with initial review group 1 or 2 in start and end cohorts.
  * Proportion of treatments with final review group 1 or 2 in start and end cohorts.
  * Distribution of indicators of change in start and end cohorts.
  * Conversion rates of review group 3a to review group 1, review group 4 to review group 1, and review group 4 to review group 3a.
  * Distribution of the reasons for the impossibility to review the target definition.
Secondary endpoints related to outcomes | 2 years
  * Toxicity [Comparison of final review groups]: Grade 3+ esophageal toxicity, Grade 3+ pulmonary toxicity (clinical and radiological), Other Grade 3+ toxicity.
  * Pattern of locoregional failure (including relation to CTV),
  * Progression free survival
  * Overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Moretti, MD, PhD, Study Chair — Belgian College of Physicians for Radiation Oncology Centers
Locations (5):
- Belgium (5):
  - GZA Ziekenhuizen (campus Sint-Augustinus), Antwerp
  - Institut Jules Bordet, Brussels
  - UZ Gent, Ghent
  - AZ Sint-Maarten, Mechelen
  - AZ Turnhout (campus Sint-Elisabeth), Turnhout

IPD SHARING:
Plan to Share IPD: No